CLINICAL TRIAL: NCT01380977
Title: Trial of Impact of Crime Group Intervention for Jail Inmates
Acronym: IOC-1
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: George Mason University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, June Tangney, Professor, George Mason University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01DA014694-1; R01DA014694 (NIH)
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Crime; Substance Abuse; HIV Risk; Criminogenic Thinking; Shame
Keywords: crime; substance abuse; HIV risk; criminogenic thinking; shame; guilt; restorative justice; victim impact group
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Impact of Crime group intervention (Experimental)
  Interventions: Behavioral: Impact of Crime group intervention
- Treatment as usual (Active Comparator)
  Interventions: Behavioral: Impact of Crime group intervention

INTERVENTIONS:
Behavioral: Impact of Crime group intervention — A group intervention for 16 1.5 hr sessions held twice a week

SUMMARY:
This pilot study is designed to evaluate the efficacy of the Impact of Crime (IOC) group intervention for jail inmates. The hypothesis is that participants in IOC will show decreases in criminogenic thinking, decreases in shame, increases in guilt, and increases in empathy, which in turn will be reflected in reduced recidivism (official records and self report), relative to those randomly assigned to a treatment as usual group.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older
* Must be male
* Must be currently incarcerated jail inmate
* Must be sentenced
* Must speak, read, and write in English with sufficient proficiency to use workbook and participate in group sessions
* Must be assigned to the jail's "general population"

Exclusion Criteria:

* Actively psychotic
* Assigned "keep separate" from other group members

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2002-08; Primary Completion 2013-08 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Self reported recidivism (arrests and undetected offenses) | 1 year post-release up to 2 yrs post release
Self reported recidivism (arrests and undetected offenses) | 4 years post-release up to 5 yrs post release
Self reported recidivism (arrests and undetected offenses) | 7 years post-release up to 8 yrs post-release
Self reported recidivism (arrests and undetected offenses) | 10 years post-release up to 11 yrs post-release
Self-reported Substance Use and Dependence - TCU | 1 year post-release up to 2 yrs post-release
Self-reported Substance Use and Dependence - TCU | 4 years post-release up to 5 yrs post-release
Self-reported Substance Use and Dependence - TCU | 7 years post-release up to 8 yrs post-release
Self-reported Substance Use and Dependence - TCU | 10 years post-release up to 11 yrs post release
Self-reported HIV risk behaviors (sex and IDU) - TCU | 1 year post-release - up to 2 yrs post-release
Self-reported HIV risk behaviors (sex and IDU) - TCU | 4 years post-release up to 5 yrs post-release
Self-reported HIV risk behaviors (sex and IDU) - TCU | 7 years post-release up to 8 yrs post-release
Self-reported HIV risk behaviors (sex and IDU) - TCU | 10 years post-release up to 11 yrs post-release

SECONDARY OUTCOMES:
Changes from baseline in Self reported criminogenic beliefs - CCS | Baseline to post-treatment up to 9 mos
Changes from baseline in Self reported criminogenic beliefs - CCS | Baseline to pre-release up to 1.5 yrs
Changes from baseline in Self reported criminogenic beliefs - CCS | Baseline to 1 yr post-release up to 3.5 yrs
Changes from baseline in Self reported criminogenic beliefs - CCS | Baseline to 4 yrs post-release up to 6.5 yrs
Changes from baseline in Self reported criminogenic beliefs - CCS | Baseline to 7 yrs post-release up 9,5 yrs
Changes from baseline in Self reported criminogenic beliefs - CCS | Baseline to 10 yrs post-release up to 12.5 yrs
Changes from baseline in self-reported shame - TOSCA-SD | Baseline to post-treatment up to 9 mos
Changes from baseline in self-reported shame - TOSCA-SD | Baseline to pre-release up to 1.5 yrs
Changes from baseline in self-reported shame - TOSCA-SD | Baseline to 1 yr post release up to 3.5 yrs
Changes from baseline in self-reported shame - TOSCA-SD | Baseline to 4 yrs post release up to 6.5 yrs
Changes from baseline in self-reported shame - TOSCA-SD | Baseline to 7 yrs post release up to 9.5 yrs
Changes from baseline in self-reported shame - TOSCA-SD | Baseline to 10 yrs post release up to 12.5 yrs
Changes from baseline in self-reported Guilt - TOSCA-SD | Baseline to post-treatment up to 9 mos
Changes from baseline in self-reported Guilt - TOSCA-SD | Baseline to pre-release up to 1.5 yrs
Changes from baseline in self-reported Guilt - TOSCA-SD | Baseline to 1 yr post-release up to 3.5 yrs
Changes from baseline in self-reported Guilt - TOSCA-SD | Baseline to 4 yrs post-release up to 6.5 yrs
Changes from baseline in self-reported Guilt - TOSCA-SD | Baseline to 7 yrs post-release up to 9.5 yrs
Changes from baseline in self-reported Guilt - TOSCA-SD | Baseline to 10 yrs post-release up to 12.5 yrs
Changes from baseline in self-reported Empathy - IRI | Baseline to post-treatment up to 9 mos
Changes from baseline in self-reported Empathy - IRI | Baseline to pre-release up to 1.5 yrs
Changes from baseline in self-reported Empathy - IRI | Baseline to 1 year post-release up to 3.5 yrs
Changes from baseline in self-reported Empathy - IRI | Baseline to 4 years post-release up to 6.5 yrs
Changes from baseline in self-reported Empathy - IRI | Baseline to 7 years post-release up to 9.5 yrs
Changes from baseline in self-reported Empathy - IRI | Baseline to 10 years post-release up to 12.5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: June P Tangney, Ph.D., Principal Investigator — George Mason University
Locations (1):
- Fairfax County Adult Detention Center, Fairfax, Virginia, United States